CLINICAL TRIAL: NCT00483366
Title: Phase I Study of Imatinib, Gemcitabine and Capecitabine in Patients With Solid Tumors
Brief Title: Imatinib Mesylate, Gemcitabine, and Capecitabine in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0163-06-FB; P30CA036727 (NIH)
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Capecitabine; Gemcitabine; Imatinib Mesylate; Base Sequence; Polymerase Chain Reaction

ARMS (1):
- Imatinib/Gemcitabine/Capecitabine (Other): Patients will be accrued on cohorts of three per dose level starting at dose level 0. Accrual to higher dose levels will depend on toxicity occurrence.
  Dose limiting toxicity (DLT) will be determined after cycle two for each patient.
  Schema: Imatinib days 1 - 5 and days 8 - 12 Gemcitabine on days 3 and 10 Capecitabine on days 1 - 14
  Doses: Imatinib 400 mg/d fixed dose Gemcitabine 450 mg/m2; 550 mg/m2; 675 mg/m2; 825 mg/m2; 1000 mg/m2 Capecitabine 500 mg/m2; 600 mg/m2 bid; 725 mg/m2; 850 mg/m2
  Treatment cycle: 21-days
  Treatment duration: Until disease progression or unacceptable toxicity defined in protocol.
  Interventions: Drug: capecitabine; Drug: gemcitabine hydrochloride; Drug: imatinib mesylate; Genetic: mutation analysis; Genetic: nucleic acid sequencing; Genetic: polymerase chain reaction

INTERVENTIONS:
Drug: capecitabine — Dose level Capecitabine
  -1 400 mg/m2 bid
  0 500 mg/m2 bid
  1. 500 mg/m2 bid
  2. 600 mg/m2 bid
  3. 600 mg/m2 bid
  4. 725 mg/m2 bid
  5. 725 mg/m2 bid
  6. 850 mg/m2 bid
  7. 850 mg/m2 bid
  Other Names: Xeloda
Drug: gemcitabine hydrochloride — Dose level Gemcitabine
  -1 400 mg/m2 0 450 mg/m2
  1. 550 mg/m2
  2. 550 mg/m2
  3. 675 mg/m2
  4. 675 mg/m2
  5. 825 mg/m2
  6. 825 mg/m2
  7. 1000 mg/m2
  Other Names: Gemzar
Drug: imatinib mesylate — Dose level Imatinib
  -1 400 mg/d 0 400 mg/d
  1. 400 mg/d
  2. 400 mg/d
  3. 400 mg/d
  4. 400 mg/d
  5. 400 mg/d
  6. 400 mg/d
  7. 400 mg/d
  Other Names: Gleevec
Genetic: mutation analysis — C-kit mutations will be assessed on existing paraffin-embedded blocks by Polymerase Chain Reaction and direct sequencing of both juxtamembrane domains (exons 9 and 11) and the tyrosine kinase domain (exons 13 and 17). Every ABI sequence will be compared to a NCBI Human KIT gene nucleotide sequence and will be blast using a NCBI Standard Nucleotide Blast Search to determine the presence of mutation within a particular exon.
Genetic: nucleic acid sequencing — C-kit mutations will be assessed on existing paraffin-embedded blocks by Polymerase Chain Reaction and direct sequencing of both juxtamembrane domains (exons 9 and 11) and the tyrosine kinase domain (exons 13 and 17). Every ABI sequence will be compared to a NCBI Human KIT gene nucleotide sequence and will be blast using a NCBI Standard Nucleotide Blast Search to determine the presence of mutation within a particular exon.
Genetic: polymerase chain reaction — C-kit mutations will be assessed on existing paraffin-embedded blocks by Polymerase Chain Reaction and direct sequencing of both juxtamembrane domains (exons 9 and 11) and the tyrosine kinase domain (exons 13 and 17). Every ABI sequence will be compared to a NCBI Human KIT gene nucleotide sequence and will be blast using a NCBI Standard Nucleotide Blast Search to determine the presence of mutation within a particular exon.

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving imatinib mesylate together with gemcitabine and capecitabine may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of gemcitabine and capecitabine when given together with imatinib mesylate in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of gemcitabine hydrochloride and capecitabine when combined with imatinib mesylate in patients with advanced solid tumors.
* Determine the toxicity of this regimen in these patients.

Secondary

* Explore the antitumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of gemcitabine and capecitabine.

Patients receive oral imatinib mesylate once daily on days 1-5 and 8-12, gemcitabine hydrochloride IV on days 3 and 10, and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days for at least 2 courses in the absence of progressive disease or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gemcitabine hydrochloride and capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Existing paraffin-embedded tissue blocks from patients diagnosed with melanoma or renal cell carcinoma will be assessed for c-kit mutations by polymerase chain reaction and direct sequencing of both juxtamembrane domains (exons 9 and 11) and tyrosine kinase domain (exon 13 and 17). (Begins 12-11-2008)

PROJECTED ACCRUAL: Closed to patient accrual 12/11/2008.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor, meeting 1 of the following criteria:

  * Failed standard therapy and subsequent line therapy
  * Disease for which no standard therapy exists
* Any number of prior therapies are allowed provided standard treatment options have either been exhausted or are unable to be administered, in the opinion of the treating physician
* Measurable or nonmeasurable disease

  * Measurable disease is defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by CT scan or ≥ 10 mm by spiral CT scan
  * Nonmeasurable disease is defined as all other lesions, including small lesions (< 20 mm by conventional techniques or < 10 mm by spiral CT scan) and truly nonmeasurable lesions, including the following:

    1. Leptomeningeal disease
    2. Bone lesions
    3. Ascites
    4. Pleural or pericardial effusion
    5. Lymphangitis cutis/pulmonis
    6. Abdominal masses that are not confirmed and followed by imaging techniques
    7. Cystic lesions
* Brain metastases allowed provided both of the following are true:

  * Patient has undergone resection and/or radiotherapy and does not require steroids
  * No evidence of disease progression by CT scan or MRI at least 4 weeks after completion of steroids, surgery, and/or radiotherapy
* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.5 g/dL (epoetin alfa supplementation allowed)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) (except if due to Gilbert's syndrome)
* AST and ALT ≤ 2.5 times ULN
* Creatinine < 1.5 times ULN
* Fertile patients must use effective barrier method contraception during and for 3 months after completion of study treatment
* Must be able to tolerate oral intake for the administration of imatinib mesylate and capecitabine
* Prior treatment with gemcitabine hydrochloride, capecitabine, or imatinib mesylate allowed provided all three drugs were not used in combination simultaneously
* Prior radiotherapy allowed provided the lesion treated is not used to assess response and has not demonstrated progression after treatment
* At least 2 weeks since prior radiotherapy
* More than 2 weeks since prior major surgery
* At least 4 weeks since prior systemic therapy (6 weeks for nitrosoureas) and recovered
* More than 4 weeks since prior packed red blood cell transfusions
* Concurrent bisphosphonate therapy allowed for skeletal metastases provided therapy is started before study entry

Exclusion Criteria:

* Not pregnant or nursing/negative pregnancy test
* No active serious infections
* No known allergy or hypersensitivity to study drugs or their formulation
* No comorbidity or condition which would preclude study participation
* No other primary malignancy within the past 5 years except basal cell skin cancer, cervical carcinoma in situ, or another primary malignancy that is not currently clinically significant or requires active intervention
* No prior radiotherapy to ≥ 25% of the bone marrow
* No concurrent anticoagulation therapy with warfarin

  * Therapeutic anticoagulation with low-molecular weight heparin or heparin allowed
  * Mini-dose warfarin (e.g., 1 mg/day) for prophylaxis of central venous catheter thrombosis allowed at the discretion of the treating physician
* No other concurrent anticancer agents, including chemotherapy and biologic agents
* No other concurrent investigational drugs
* No concurrent routine systemic corticosteroid therapy (corticosteroid therapy may only be administered after consultation with the principal investigator)
* No other malignant disease
* No New York Heart Association class III-IV cardiac disease
* No congestive heart failure
* No myocardial infarction within the past 6 months
* No known chronic liver disease (e.g., chronic active hepatitis or cirrhosis)
* No known HIV infection
* No prior radiotherapy to ≥ 25% of the bone marrow
* No concurrent anticoagulation therapy with warfarin

  * Therapeutic anticoagulation with low-molecular weight heparin or heparin allowed
  * Mini-dose warfarin (e.g., 1 mg/day) for prophylaxis of central venous catheter thrombosis allowed at the discretion of the treating physician
* No other concurrent anticancer agents, including chemotherapy and biologic agents
* No other concurrent investigational drugs
* No concurrent routine systemic corticosteroid therapy (corticosteroid therapy may only be administered after consultation with the principal investigator)

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-08-15 (Actual); Primary Completion 2009-01-30 (Actual); Study Completion 2011-03-29 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of gemcitabine hydrochloride and capecitabine when combined with imatinib mesylate | By the end of cycle 2
  Cohorts of 3 starting at dose level 0. The imatinib dose is fixed. The dose of capecitabine is initially fixed and the dose of gemcitabine is increased 1 dose level. For the subsequent cohort, the dose of gemcitabine will be fixed and the dose of capecitabine advanced to the next dose level. 3 patients will be treated on the initial schedule. If no dose-limiting toxicities related to drug are observed and no patients require dose mods by the end of cycle 2, then 3 patients will be treated on the next schedule.
Dose-limiting Toxicity | By the end of cycle 2.
  Cohorts of 3 starting at dose level 0. The imatinib dose is fixed. The dose of capecitabine is initially fixed and the dose of gemcitabine is increased 1 dose level. For the subsequent cohort, the dose of gemcitabine will be fixed and the dose of capecitabine advanced to the next dose level. 3 patients will be treated on the initial schedule. If no dose-limiting toxicities related to drug are observed and no patients require dose mods by the end of cycle 2, then 3 patients will be treated on the next schedule.

SECONDARY OUTCOMES:
Antitumor activity | Following response assessment.
  Deidentified melanoma samples will be sent to our collaborator at Ohio State, Dr. Christopher Corless, who is a recognized expert in this field. Renal cell samples will be assayed here at our institution

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Hauke, MD, Principal Investigator — University of Nebraska; Elizabeth C. Reed, MD, Study Chair — University of Nebraska
Locations (1):
- UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska, United States